CLINICAL TRIAL: NCT07403656
Title: Acil Servis Hemşirelerin Deneyimledikleri Travma ve Rutin Stresörlerin İncelenmesi
Brief Title: Traumatic and Routine Stressors Experienced by Emergency Nurses
Acronym: TRSS-ED
Status: Completed | Type: Observational
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Department of Nursing, Agri Ibrahim Cecen University
Other Study IDs: AICU-TRSS-ED-2025
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Occupational Stress; Work-Related Psychological Stress; Traumatic Stress; Burnout, Psychological
Keywords: Emergency Nurses; Traumatic and Routine Stressors; Occupational Stress; Emotional Impact; Emergency Department; Mental Health; Cross-Sectional Study
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological; Emergencies; Psychological Well-Being | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency Nurses: Registered nurses working in emergency departments who participated in this observational, cross-sectional study.
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — This study is observational and does not involve any intervention. Participants completed self-administered questionnaires only.

SUMMARY:
Emergency nurses are frequently exposed to both traumatic events and routine work-related stressors due to the nature of emergency care settings. These experiences may have important emotional and psychological effects, which can influence nurses' well-being, job satisfaction, and quality of patient care.

The aim of this study is to examine the frequency and emotional impact of traumatic and routine stressors experienced by emergency department nurses during the past six months. The study focuses on identifying common stressors and understanding how often these events occur and how strongly they affect nurses emotionally.

This observational, cross-sectional study was conducted among emergency nurses working in public hospitals in Turkey. Data were collected using a structured questionnaire that includes demographic questions and the Traumatic and Routine Stressors Scale (TRSS-TR), a validated instrument designed specifically for emergency nurses.

The findings of this study are expected to contribute to a better understanding of occupational stress among emergency nurses and to support the development of strategies aimed at protecting nurses' mental health and improving working conditions in emergency care environments.

DETAILED DESCRIPTION:
Emergency departments are high-intensity clinical environments where nurses are regularly exposed to traumatic events such as sudden death, severe injuries, violence, and resuscitation efforts, as well as routine stressors including high workload, time pressure, communication challenges with patients' relatives, and limitations in providing optimal care. While traumatic events are often sudden and emotionally intense, routine stressors may appear less severe but can accumulate over time and lead to significant psychological burden.

This study was designed as an observational, descriptive, and cross-sectional investigation to systematically examine both traumatic and routine stressors experienced by emergency department nurses and to evaluate the emotional impact of these experiences. The study was conducted in multiple public hospitals located in different regions of Turkey, reflecting the multi-center nature of emergency nursing practice.

The study population consisted of registered nurses working in emergency departments. Eligibility criteria included having at least six months of experience in an emergency department and voluntary agreement to participate in the study. Nurses who met these criteria were invited to complete an anonymous, self-administered online questionnaire.

Data collection took place between September 1, 2025, and December 1, 2025. The questionnaire included two main components: a demographic information form and the Traumatic and Routine Stressors Scale - Turkish Version (TRSS-TR). The TRSS-TR is a validated and reliable instrument adapted for use among Turkish emergency nurses. The scale assesses both the frequency of exposure to specific traumatic and routine stressors during the past six months and the perceived emotional impact of each stressor. Responses are rated on Likert-type scales, allowing for quantitative analysis of stressor exposure and emotional burden.

All data were collected anonymously using a secure online survey platform. Participation was entirely voluntary, and informed consent was obtained electronically from all participants prior to data collection. No identifying personal information was collected.

Data analysis was performed using statistical software. Descriptive statistics were used to summarize demographic characteristics and scale scores. Depending on data distribution, appropriate parametric or non-parametric tests were applied to examine relationships between stressor frequency, emotional impact, and selected demographic or occupational variables. Statistical significance was set at p < 0.05.

This study does not involve any intervention, experimental treatment, drug, or medical device. There are no anticipated physical or clinical risks to participants. The study protocol was reviewed and approved by the Ethics Committee of Agri Ibrahim Cecen University. The results are expected to provide evidence-based insights into occupational stress among emergency nurses and to inform future initiatives aimed at improving mental health support, workplace resilience, and organizational policies in emergency care settings.

ELIGIBILITY:
* Inclusion Criteria;
* Registered nurses working in emergency departments
* At least 6 months of experience working in an emergency department
* Aged 18 years or older
* Willingness to participate voluntarily in the study
* Ability to complete an online self-administered questionnaire
* Exclusion Criteria ;
* Less than 6 months of experience working in an emergency department
* Refusal or inability to provide informed consent
* Incomplete questionnaire responses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of registered nurses working in emergency departments of public hospitals in Turkey. Participants are adult nurses with at least six months of emergency department experience who voluntarily agreed to participate in this observational, cross-sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Frequency and Emotional Impact Scores of Traumatic and Routine Stressors | One-time assessment covering stressor exposure and emotional impact over the previous 6 months
  The primary outcome is the frequency and emotional impact of traumatic and routine stressors experienced by emergency department nurses, measured using the Traumatic and Routine Stressors Scale - Turkish Version (TRSS-TR).
  The frequency subscale assesses how often each stressor was experienced during the past six months using a 7-point Likert scale ranging from 1 ("less than three times in six months") to 7 ("daily"). The emotional impact subscale evaluates the perceived emotional impact of each stressor using a 7-point Likert scale ranging from 1 ("no emotional impact") to 7 ("maximum emotional impact").
  Outcome measures are reported as continuous scale scores for frequency and emotional impact, with higher scores indicating greater exposure frequency and higher perceived emotional impact.

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Dr. Murat Dilmener Training and Research Hospital, Istanbul, Bostancı
  - Dogubayazit State Hospital, Ağrı, Dogubeyazit
  - Ağrı Training and Research Hospital, Ağrı, Merkez
  - Taksim Training and Research Hospital, Istanbul, Taksim

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves anonymous self-reported questionnaire data collected from healthcare professionals and includes sensitive occupational and psychological information. Data sharing was not included in the original ethics committee approval, and therefore individual-level data will be used only for the purposes of this study and related scientific publications.

REFERENCES:
- [Background] Hetherington D, Wilson NJ, Dixon K, Murphy G. Emergency department Nurses' narratives of burnout: Changing roles and boundaries. Int Emerg Nurs. 2024 Jun;74:101439. doi: 10.1016/j.ienj.2024.101439. Epub 2024 Apr 5. PMID 38581856
- [Background] PMID: 38374938
- [Background] McCormick E, Devine S, Crilly J, Brough P, Greenslade J. Measuring occupational stress in emergency departments. Emerg Med Australas. 2023 Apr;35(2):234-241. doi: 10.1111/1742-6723.14101. Epub 2022 Oct 25. PMID 36283708
- [Background] Mirzaei A, Mozaffari N, Habibi Soola A. Occupational stress and its relationship with spiritual coping among emergency department nurses and emergency medical services staff. Int Emerg Nurs. 2022 May;62:101170. doi: 10.1016/j.ienj.2022.101170. Epub 2022 Apr 26. PMID 35487041
- [Background] Gomez-Urquiza JL, De la Fuente-Solana EI, Albendin-Garcia L, Vargas-Pecino C, Ortega-Campos EM, Canadas-De la Fuente GA. Prevalence of Burnout Syndrome in Emergency Nurses: A Meta-Analysis. Crit Care Nurse. 2017 Oct;37(5):e1-e9. doi: 10.4037/ccn2017508. PMID 28966203